CLINICAL TRIAL: NCT04358237
Title: Phase I/II, Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination With Pembrolizumab in Patients With Relapsed Small Cell Lung Cancer
Brief Title: Lurbinectedin (PM01183) Combined With Pembrolizumab in Small Cell Lung Cancer.
Acronym: LUPER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antonio Calles Blanco (Other)
Collaborators: MedSIR (Other); PharmaMar (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Antonio Calles Blanco, Physician Thoracic Oncology, Head & Neck and Sarcoma Unit Early Drug Development and Phase I Unit, Blanco, Dr Antonio Calles MD
Organization: Blanco, Dr Antonio Calles MD (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP300
Record Dates: First submitted 2020-04-03; First posted 2020-04-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Relapsed
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — PM 01183; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase I/II, Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination with Pembrolizumab in Patients with Relapsed Small Cell Lung Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: lurbinectedin (PM01183) + pembrolizumab (Experimental): During the phase I stage, patients will start receiving pembrolizumab at a fixed dose of 200 mg as a 30-min intravenous (IV) infusion followed by lurbinectedin at a starting dose of 2.4 mg/m2 as a 1-h IV infusion on Day 1, both every 3 weeks (Q3W). Lurbinectedin dose will be escalated from the starting dose in successive cohorts of patients, with a pre-established fixed dose increase (in mg/m2) of approximately 30%.
  During the phase II stage, patients will receive pembrolizumab at a fixed dose of 200 mg as a 30-min IV infusion followed by lurbinectedin as a 1-h IV infusion on Day 1 Q3W at the redommended dose (RD) determined during the phase I stage. A cycle is defined as an interval of 3 weeks. No dose escalation will be allowed during the phase II stage.
  Interventions: Drug: Lurbinectedin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lurbinectedin — Lurbinectedin will be presented as a lyophilized powder for concentrate for solution for infusion in 4-mg vials. Before use, the 4-mg vial will be reconstituted with 8 mL of sterile water for injection, to give a solution containing 0.5 mg/mL of PM01183. For administration to patients as IV infusion, reconstituted vials will be diluted with glucose 50 mg/mL (5%) or sodium chloride 9 mg/mL (0.9%) solution for infusion.
  PM01183 will be administered as a 1 hour IV infusion Q3W, in a minimum volume of 100 mL of solution for infusion (either 5% glucose or 0.9% sodium chloride), or a minimum volume of 250 mL if through a peripheral line, always at a fixed rate and through a pump device.
  Other Names: PM01183; Zepsyre
Drug: Pembrolizumab — Pembrolizumab will be supplied as a solution for infusion in a single-use vial. Each vial contains 100 mg of MK3475 (pembrolizumab) in 4 ml of solution. Pembrolizumab 200 mg will be administered as a 30 minute IV infusion Q3W.
  Other Names: Keytruda

SUMMARY:
This is a prospective, open-label, uncontrolled and multicenter phase I/II study of PM01183 in combination with pembrolizumab in patients with relapsed small cell lung cancer (SCLC).

The study will be divided into two stages:

* A dose-ranging phase I stage with escalating doses of PM01183 in combination with a fixed dose of pembrolizumab, followed by:
* A non-randomized phase II stage as an expansion study at the recommended dose (RD) determined during the phase I stage.

The phase I stage will focus on the selection of the RD based on safety/tolerability, while the phase II stage will assess the overall response rate (ORR) and clinical response.

DETAILED DESCRIPTION:
• During the phase I stage, patients will start receiving pembrolizumab at a fixed dose of 200 mg as a 30-min intravenous (IV) infusion followed by PM01183 at a starting dose of 2.4 mg/m2 as a 1-h IV infusion on Day 1, both every 3 weeks (Q3W). A cycle is defined as an interval of 3 weeks.

PM01183 dose will be escalated from the starting dose in successive cohorts of patients, with a pre-established fixed dose increase (in mg/m2) of approximately 30%.

Dose escalation will follow a classical 3+3 design, according to the observed tolerance and safety. All evaluable patients within a dose level will be followed for at least one cycle (i.e., 3 weeks) before dose escalation may proceed. The maximum tolerated dose (MTD) will be the lowest dose level explored during dose escalation at which one third or more of evaluable patients experience a dose-limiting toxicity (DLT) in Cycle 1.

Dose escalation will be terminated once the MTD or the last dose level (i.e., DL2) is reached, whichever occurs first, except if all DLTs occurring at a given dose level are related to neutropenia. If this is the case, dose escalation may be resumed, starting at the lowest dose level at which exclusively neutropenia-related DLTs were observed, and will follow the same original schedule but with mandatory primary granulocyte colony-stimulating factor (G-CSF) prophylaxis.

An expansion cohort to complete a minimum of 6 evaluable patients will be recruited at the immediate lower dose level from the MTD, or at DL2 if the MTD is not defined yet. This level will be confirmed as the RD if less than one third of the first 6 evaluable patients experience DLT during Cycle 1. Intermediate dose levels could be tested upon agreement of the Scientific Steering Committee members, as defined in Section 8.4, if deemed appropriate. This will also be discussed with Pharma Mar and MSD.

• During the phase II stage, patients will receive pembrolizumab at a fixed dose of 200 mg as a 30-min IV infusion followed by PM01183 as a 1-h IV infusion on Day 1 Q3W at the RD determined during the phase I stage. A cycle is defined as an interval of 3 weeks. No dose escalation will be allowed during the phase II stage.

Regardless of stage, patients will receive PM01183 in combination with pembrolizumab until progression, unacceptable toxicity, consent withdrawal or if it is not considered in their best interest to continue, after specific agreement between the Investigators and the Sponsor (this will also be discussed with Pharma Mar and MSD). Maximum treatment period with pembrolizumab is 35 dose administrations (approximately 2 years). After 35 dose administrations, patients might continue on treatment with lurbinectedin alone.

Radiological tumor assessments will be done every 6 weeks (± 2 weeks), or prior to every second subsequent cycle, while on treatment. After treatment discontinuation, patients will be followed until resolution or stabilization of all toxicities, if any. Patients discontinuing treatment without disease progression as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 will be followed every 6 weeks (± 2 weeks) until disease progression as per RECIST 1.1, start of a new anti-cancer therapy, death or the end-of-study date (clinical cutoff, as described in Section 2.1.1), whichever occurs first. After one year of follow-up, patients will be evaluated every 9 weeks (± 2 weeks) until the end of the study.

After disease progression as per RECIST 1.1 or start of a new anti-cancer therapy, patients will be followed up for survival every 12 weeks (± 2 weeks) until death or the end-of-study date, whichever occurs first (a phone contact will be acceptable). An exception will be those patients who are clinically stable at the time of disease progression as per RECIST 1.1, who could remain on treatment according to the Investigator's criteria up to the next radiological assessment. If no disease progression as per immune RECIST (iRECIST) 1.1 is observed in this assessment, treatment will continue until disease progression as per iRECIST 1.1.

If at the end of the study (i.e., clinical cut-off, as defined in Section 2.1.1) any patients are still on treatment with lurbinectedin monotherapy, the investigator will evaluate if it is appropriate that they continue receiving that treatment. If needed, the Sponsor may facilitate appropriate measures to ensure access to lurbinectedin and maintenance of safety reporting obligations beyond study closure in those cases. According to the end of study definition (see Section 2.1.1), no patients will remain under treatment with pembrolizumab at the clinical cut-off.

Safety will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5, whereas antitumor response will be assessed using the RECIST 1.1, and also the iRECIST 1.1 whenever applicable. These methods are generally accepted as standard clinical procedures in oncological studies.

ELIGIBILITY:
Inclusion criteria

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of SCLC whose disease has progressed after first-line chemotherapy-based regimen will be enrolled in this study.
2. At least 4 weeks since the last anticancer therapy.
3. Male participants: a male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 190 days after the last dose of study treatment and refrain from donating sperm during this period.
4. Female participants: a female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 7 months after the last dose of study treatment.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1. Evaluation of ECOG PS is to be performed within 7 days prior to the date of allocation.
8. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.
9. Recovery to NCI-CTCAE grade ≤1 or to baseline from any AE derived from previous treatment (excluding alopecia and/or cutaneous toxicity and/or peripheral sensory neuropathy and/or asthenia, all grade ≤2 and/or correctable electrolyte abnormality with supplementation).
10. Patients included in the expansion cohort at the RD (stage I) and all patients included in the stage II must have:

    1. Measurable disease according to RECIST 1.1; and
    2. Documented disease progression during or immediately after last therapy according to any of the aforementioned criteria.

Exclusion criteria

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has had prior treatment with or exposure to: a) PM01183. b) T-cell or other cell-based or biologic therapies. c) Experimental anti-tumor vaccines; therapies that target any T-cell co- stimulation or checkpoint pathways, such as anti-PD-1, anti-PD-L1, anti-PD- L2, anti-CD137, or anti CTLA-4 antibody, including ipilimumab; or other medicines specifically targeting T-cells.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has had radiotherapy (RT) in more than 35% of the bone marrow.
6. Has a history of previous bone marrow and/or stem cell transplantation and allogenic transplant.
7. Has an impending need for RT (e.g., painful bone metastasis and/or risk of spinal cord compression).
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
9. Has any of the following concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
   2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
   3. History of idiopathic, pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis or evidence of active pneumonitis on screening chest CT-scan. History of radiation pneumonitis in radiation field (fibrosis) is permitted, as long as it is asymptomatic and no steroids are needed.
   4. Known history of active neurologic paraneoplastic syndrome.
   5. Myopathy or any clinical situation that causes significant and persistent elevation of CPK (>2.5 x ULN in two different determinations performed one week apart).
   6. Limitation of the patient's ability to comply with the treatment or follow-up protocol.
   7. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
13. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment. Brain CT-scan or MRI results must be provided at baseline.
14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, PM01183 and/or any of their excipients.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Exception: patients with vitiligo or resolved childhood asthma/atopy; patients who require intermittent use of bronchodilators or local steroid injections; and patients with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.
16. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
17. Has an active infection requiring systemic therapy.
18. Has a known history of Human Immunodeficiency Virus (HIV).
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
20. Has a known history of active tuberculosis (Mycobacterium tuberculosis).
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) and recommended phase II dose (RD) of lurbinectedin in combination with pembrolizumab in patients with relapsed SCLC. | 12 months
  The MTD will be the lowest dose level explored during dose escalation at which more than one third of evaluable patients develop a DLT in Cycle 1. The RD will be the highest dose level explored at which less than one third of evaluable patients develop a DLT during Cycle 1.
Phase II: Efficacy of lurbinectedin in combination with pembrolizumab in terms of overall response rate (ORR), according to RECIST 1.1, in patients with relapsed SCLC. | 38 months
  ORR is defined as the percentage of evaluable patients with a confirmed response, either complete (CR) or partial (PR).
  The ORR will be assessed using the RECIST 1.1 on a set of measurable lesions identified at baseline as target lesions or as non-target lesions (if any), and followed until PD by an appropriate method.

SECONDARY OUTCOMES:
Phase I: Preliminary information on the clinical antitumor activity of the combination. | 28 months
  Preliminary antitumor activity in the phase I stage will be evaluated according to the RECIST 1.1 (and the iRECIST 1.1, whenever applicable) at least 6 weeks after treatment initiation in all patients with measurable disease.
Phase I: MTD and RD of lurbinectedin in combination with pembrolizumab with mandatory primary prophylaxis with G-CSF in patients with relapsed SCLC (if DLTs of this combination are exclusively related to neutropenia). | 12 months
  The MTD will be the lowest dose level explored during dose escalation at which more than one third of evaluable patients develop a DLT in Cycle 1. The RD will be the highest dose level explored at which less than one third of evaluable patients develop a DLT during Cycle 1.
Phase II: Antitumor activity of this combination as per RECIST 1.1 (and iRECIST 1.1, whenever applicable) in terms of Clinical benefit ≥3 months. | 38 months
  During expansion at the RD in the phase II stage, antitumor activity will also be evaluated according to the RECIST 1.1 (and the iRECIST 1.1, whenever applicable).
Phase II: Antitumor activity of this combination as per RECIST 1.1 (and iRECIST 1.1, whenever applicable) in terms of Duration of response (DOR). | 38 months
  During expansion at the RD in the phase II stage, antitumor activity will also be evaluated according to the RECIST 1.1 (and the iRECIST 1.1, whenever applicable).
Phase II: Antitumor activity of this combination as per RECIST 1.1 (and iRECIST 1.1, whenever applicable) in terms of Progression-free survival (PFS). | 38 months
  During expansion at the RD in the phase II stage, antitumor activity will also be evaluated according to the RECIST 1.1 (and the iRECIST 1.1, whenever applicable).
Phase II: Antitumor activity of this combination as per RECIST 1.1 (and iRECIST 1.1, whenever applicable) in terms of Overall survival (OS). | 38 months
  During expansion at the RD in the phase II stage, antitumor activity will also be evaluated according to the RECIST 1.1 (and the iRECIST 1.1, whenever applicable).
Both Stages: Safety profile and feasibility of lurbinectedin in combination with pembrolizumab in patients with relapsed SCLC. | 38 months
  Patients will be evaluable for safety if they have received at least one partial infusion of lurbinectedin. AEs will be graded according to the NCI-CTCAE v.5. Additionally, treatment compliance, in particular dose reduction requirements, skipped doses and/or cycle delays due to AEs, will be described.
Both stages: Characterize the plasma pharmacokinetics (PK) of lurbinectedin in this combination and to detect major drug-drug PK interactions. | 38 months
  PK parameters (CMax) will be evaluated in plasma by standard non-compartmental methods (compartmental modeling may be performed if appropriate).
Both stages: Pharmacogenetic (PGt) analysis. | 38 months
  A blood sample will be collected at any time during the trial (but preferably just before treatment start in Cycle 1 along with the first PK sample) to analyze germline DNA for the presence or absence of mutations or polymorphisms in genes relevant for the metabolism and/or transport of lurbinectedin that may help explain individual variability in main PK parameters.
Both stages: Pharmacogenomic (PGx) analysis in tumor samples of patients exposed to lurbinectedin and pembrolizumab in order to assess potential markers of response and/or resistance. | 38 months
  The mutational status of factors involved in DNA repair mechanisms, or related to the mechanism of action of PM01183 or pembrolizumab, will be evaluated from available prior paraffin-embedded tumor tissue samples obtained at diagnosis or relapse. mRNA and/or protein expression levels of these factors might be also analyzed, if relevant. Potentially whole exome sequencing will also be analyzed. Their correlation with the clinical response and outcome after treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Calles, Principal Investigator — Hospital Gregorio Marañon
Locations (5):
- Spain (5):
  - Hospital Vall D´Hebrón, Barcelona
  - ICO - Instituto Catalán de Oncología, Barcelona
  - Hospital Gregorio Marañon, Madrid
  - START - Phase I Unit - HN San Chinarro, Madrid
  - Start - Unidad Fase I - Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No